CLINICAL TRIAL: NCT01157026
Title: Effectiveness of Tocotrienol-rich Fraction Combined With Tamoxifen in the Management of Women With Early Breast Cancer: A Pilot Clinical Trial
Brief Title: A Pilot Clinical Trial With Tocotrienol on Breast Cancer
Acronym: BC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Responsible Party: Kalanithi Nesaretnam, Malaysian Palm Oil Board
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT369; 5399 S1 (Registry Identifier: National Medical Research Register,Malaysia)
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Tocotrienol-rich fraction with tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tocotrienol Rich Fraction plus Tamoxifen (Experimental)
  Interventions: Dietary Supplement: Tocotrienol Rich Fraction (TRF)
- Placebo plus tamoxifen (Active Comparator)
  Interventions: Other: placebo plus tamoxifen

INTERVENTIONS:
Dietary Supplement: Tocotrienol Rich Fraction (TRF) — Tocotrienol Rich Fraction (200mg), daily for five years
  Other Names: Tocotrienol Rich Fraction (Hovid Sdn.Bhd)
  Arms: Tocotrienol Rich Fraction plus Tamoxifen
Other: placebo plus tamoxifen — 20mg tamoxifen daily
  Arms: Placebo plus tamoxifen

SUMMARY:
Tocotrienol Rich Fraction (TRF) in combination with Tamoxifen will improve breast cancer specific survival and recurrence free survival, in women with early breast cancer and estrogen receptor positive tumors.

DETAILED DESCRIPTION:
We conducted a, double-blinded, placebo controlled trial of TRF plus tamoxifen versus placebo plus tamoxifen in women with primary breast cancer for five years. Both the TRF and placebo drugs were prepared and supplied by Hovid Sdn Bhd, Malaysia. Hovid Sdn. Bhd. absolutely did not have any influence in the trial designing, patient recruitment, data collection, analysis and reporting. The placebo drug which contained soy oil without tocotrienols had similar appearance and taste as the TRF drug. A total of 240 women breast cancer patients were assigned to two groups by minimization method that balanced treatment groups. The intervention group was given TRF plus tamoxifen, (n = 120) while control group was given placebo plus tamoxifen, (n = 120). The primary end point was breast cancer specific survival, defined as the time from minimization to death due to breast cancer. The secondary end points included disease free survival, biochemical parameters, liver function and plasma levels of vitamin E.

ELIGIBILITY:
Inclusion criteria:

1. women with estrogen receptor positive tumors.
2. 40-60 years of age at the start of the tamoxifen therapy.
3. histologically confirmed primary breast cancer.
4. a tumor that was positive for estrogen receptors, progesterone receptors, or both.
5. an Eastern Cooperative Oncology Group performance status of 0,1, or 2 (scored on a scale of 0 to 5, with lower scores indicating better function).

Exclusion criteria:

1. concurrent use of investigational drugs and estrogen receptor status negative or unknown.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2001-11; Primary Completion 2006-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
breast cancer specific survival | Five Years
  defined as the time from minimization to death due to breast cancer

SECONDARY OUTCOMES:
disease free survival | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Kalanithi Nesaretnam, PhD, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysian Palm Oil Board, Kajang, Selangor, Malaysia

REFERENCES:
- [Derived] Nesaretnam K, Selvaduray KR, Abdul Razak G, Veerasenan SD, Gomez PA. Effectiveness of tocotrienol-rich fraction combined with tamoxifen in the management of women with early breast cancer: a pilot clinical trial. Breast Cancer Res. 2010;12(5):R81. doi: 10.1186/bcr2726. Epub 2010 Oct 8. PMID 20929592